CLINICAL TRIAL: NCT02418195
Title: Plasma Exosomal MicroRNAs as Promising Novel Biomarkers for Suicidality and Treatment Outcome
Brief Title: miRNAs, Suicide, and Ketamine - Plasma Exosomal microRNAs as Novel Biomarkers for Suicidality and Treatment Outcome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yogesh Dwivedi, PhD, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: F141029007; 1R01MH107183-01 (NIH)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Ketamine; Suicide Attempt; Suicidal Ideation; Suicidality
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Suicide, Attempted; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MDD with recent Suicide Attempt (Active Comparator): All subjects with Major Depressive Disorder with a recent Suicide Attempt (in the past 2 weeks) will receive a one-time IV infusion of ketamine at a dose of 0.5mg/kg at a rate of 40 milliliters (mL) over 40 minutes. Blood will be drawn at pre-dose, 30 minutes post dose, 180 minutes post dose, 24 hours post dose, and 14 days post dose to measure changes in miRNAs.
  Interventions: Drug: ketamine
- MDD with Suicidal Ideation no attempt (Active Comparator): All subjects with Major Depressive Disorder with recent Suicidal Ideation (in the past 7 days) without a recent Suicide Attempt (in the past 6 months) will receive a one-time IV infusion of ketamine at a dose of 0.5mg/kg at a rate of 40mL over 40 minutes. Blood will be drawn at pre-dose, 30 minutes post dose, 180 minutes post dose, 24 hours post dose, and 14 days post dose to measure changes in miRNAs.
  Interventions: Drug: ketamine
- MDD without Suicidal Ideation no attempt (Active Comparator): All subjects with Major Depressive Disorder without recent Suicidal Ideation (in the past 7 days) without a recent Suicide Attempt (in the past 6 months) will receive a one-time IV infusion of ketamine at a dose of 0.5mg/kg at a rate of 40mL over 40 minutes. Blood will be drawn at pre-dose, 30 minutes post dose, 180 minutes post dose, 24 hours post dose, and 14 days post dose to measure changes in miRNAs.
  Interventions: Drug: ketamine
- Healthy Controls (No Intervention): Healthy Control subjects without a psychiatric diagnosis will have a one-time blood draw to examine miRNAs.

INTERVENTIONS:
Drug: ketamine — IV infusion of ketamine 0.5mg/kg at a rate of 40mL over 40 minutes
  Other Names: ketalar
  Arms: MDD with Suicidal Ideation no attempt; MDD with recent Suicide Attempt; MDD without Suicidal Ideation no attempt

SUMMARY:
The purpose of this study is to examine whether neural-derived exosomal miRNAs are differentially expressed that are specific to suicidal ideation or behavior, and which by affecting specific miRNA targets and pathways, are associated with suicidal behavior and response to ketamine. The following groups of subjects will be examined: 1) major depressive disorder (MDD) with a recent suicide attempt (in past 2 weeks), 2) MDD with serious ideation (in the past 7 days) without recent suicide attempt (in the past 6 months), 3) MDD without clinically significant suicidal ideation (in the past 7 days) or recent suicide attempt (in the past 6 months), and 4) healthy controls. Both suicidal and non-suicidal MDD will be given ketamine (0.5 mg/kg, IV) and blood will be drawn at predose, 30 min, 180 min, 24 hours, and 14 days post-infusion to measure changes in miRNAs.

As of May 2022, study is in data analysis. Final outcomes will be known once analysis is complete.

As of July 2022, all data collection is complete. The primary and secondary data outcome measure results are complete.

The investigators are working on final analysis of the mRNA samples, to provide final responses to questions posed in the Detailed Description section below and listed here: 1) whether suicidal ideation or behavior is associated with differences in the expression of specific miRNAs, 2) whether anti-suicidal/antidepressant effects of ketamine is associated with miRNAs changes, and 3) whether miRNA/mRNA-regulatory pathways contribute to suicide pathogenesis and treatment response.

DETAILED DESCRIPTION:
Neural MicroRNAs (miRNAs) are responsive to environmental, synaptic, and pathological changes and can be actively secreted by cells such as exosomes from brain into blood. These exosomes bear cell-type specific surface markers. Using a neural specific surface marker, the investigators successfully isolated neural-derived exosomes and found that these exosomes are enriched with miRNAs/Messenger RNA (mRNAs) that are expressed in brain. Using this novel approach the investigators aim to examine whether neural derived exosomal miRNAs are differentially expressed that are specific to suicidal ideation or behavior, and which by affecting specific mRNA targets and pathways, are associated with suicidal behavior and response to ketamine.

The following groups of subjects will be examined: 1) major depressive disorder (MDD) with a recent suicide attempt (in past 2 weeks), 2) MDD with serious ideation (in the past 7 days) without recent suicide attempt (in the past 6 months), 3) MDD without clinically significant suicidal ideation (in the past 7 days) or suicide attempt in the past 6 months, and 4) healthy controls. Both suicidal and non-suicidal MDD will be given ketamine (0.5 mg/kg, IV) and blood will be drawn at pre-infusion, 30 minutes and 180 minutes post-infusion to measure changes in miRNAs. Healthy controls will have a one-time blood draw. The investigators also propose a parallel human postmortem brain study to examine whether changes in miRNAs in suicidality correspond to miRNA changes in brain by comparing dlPFC and hippocampus from MDD suicide, MDD non-suicide, and control subjects.

With this the investigators attempt to discover 1) whether suicidal ideation or behavior is associated with differences in the expression of specific miRNAs, 2) whether anti-suicidal/antidepressant effects of ketamine is associated with miRNAs changes, and 3) whether miRNA/mRNA-regulatory pathways contribute to suicide pathogenesis and treatment response. Our study will provide a novel avenue for the development of miRNAs as ''molecular tool'' to identify suicidality and treatment response and in generating target based therapies to treat this devastating disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Physically healthy and capable of undergoing ketamine infusion
3. Willing and able to provide informed consent
4. Diagnosis of Major Depressive Episode (MDE) as determined by the Mini International Neuropsychiatric Interview (MINI) (MDD participants)
5. Hamilton Depression Rating Scale (HAM-D) 21 score ≥ 16 (MDD participants)
6. Suicide attempt occurred within past 2 weeks (MDD Participants with Suicide Attempt)
7. For the time frame of the past 7 days, Columbia-Suicide Severity Rating Scale (C-SSRS) score ≥ 3 (MDD Participants without Suicide Attempt, with Suicidal Ideation)
8. For the time frame of the past 7 days, C-SSRS score < 3 (MDD Participants without Suicide Attempt, without SUicidal Ideation)

Exclusion Criteria:

1. Pregnancy or lactation
2. Post-partum state (being within 2 months of delivery or miscarriage)
3. Homicide risk as determined by clinical interview
4. A lifetime history of psychotic disorder
5. Any history of dissociation or dissociative disorder
6. Bipolar disorder
7. Pervasive developmental disorder
8. Cognitive disorder
9. Cluster A personality disorder
10. Anorexia nervosa
11. Treatment with one of the following medications, known to affect the glutamate-N-methyl-D-aspartate (NMDA) receptor system (specifically: lamotrigine, acamprosate, memantine, riluzole, or lithium)
12. Alcohol or drug dependence (except nicotine and caffeine) within the last month or the use of any hallucinogen (except cannabis), including phencyclidine in the last month
13. Any known hypersensitivity or serious adverse effect associated with ketamine treatment
14. Any clinically-significant medication condition or therapy that would preclude treatment with ketamine, to include: Recent myocardial infarction
15. Unstable angina
16. Active neoplasm in the past 6 months
17. Immunosuppressive or corticosteroid therapy within the last month, with the following exceptions: any inhaled, intranasal, topical or vaginal corticosteroids are allowed.
18. Chemotherapy
19. Head injury of loss of consciousness in the past 6 months
20. If the subject reports any of the following disorders:

    * Rheumatoid arthritis
    * Lupus erythematosus
    * Autoimmune hepatitis
    * Autoimmune peripheral neuropathy
    * Autoimmune pancreatitis
    * Behcet's disease
    * Chrohn's disease
    * Autoimmune glomerulonephritis
    * Grave's disease
    * Guillain-Barre syndrome (if active)
    * Hashimoto's thyroiditis
    * Autoimmune polymyositis or polymyalgia (fibromyalgia is OK)
    * Myasthenia gravis
    * Narcolepsy
    * Polyarteritis nodosa
    * Scleroderma
    * Sjogren's syndrome
    * Transverse myelitis
    * Wegener's granulomatosis
    * HIstory of seizures (only childhood febrile seizures allowed)
    * (HIV and Hepatitis are OK if stable)
21. Systolic blood pressure > 150 and/or diastolic blood pressure >90 at screening
22. A Corrected QT Interval (QTc) > 480 msec as determined by an ECG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Dwivedi, Ph.D., Principal Investigator — University of Alabama at Birmingham; Richard C Shelton, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled April 2015 through December 2020. The last subject completed their final visit on December 30, 2020. Participants were enrolled through advertising means, such as flyers, physician referrals, sub-I clinic referrals, and chart review, via Impact.
  As of May 2022, study is in data analysis. Final outcomes will be known once analysis is complete.
Pre-assignment Details: A number of participants were excluded for not meeting inclusion or meeting exclusion criteria, in total 51. These were considered screen failures.
Period: Overall Study
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt | Healthy Controls
Started | 62 (Number subjects screened in this group.) | 63 (Number subjects screened in this group.) | 61 (Number subjects screened in this group.) | 61 (Number subjects screened in this group.)
Completed | 62 (Number subjects screened in this group.) | 63 (Number subjects screened in this group.) | 61 (Number subjects screened in this group.) | 61 (Number subjects screened in this group.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MDD With Recent Suicide Attempt: All subjects with Major Depressive Disorder with a recent Suicide Attempt (in the past 2 weeks) will receive a one-time IV infusion of ketamine at a dose of 0.5mg/kg at a rate of 40mL over 40 minutes. Blood will be drawn at pre-dose, 30 minutes post dose, 180 minutes post dose, 24 hours post dose, and 14 days post dose to measure changes in miRNAs.
  ketamine: IV infusion of ketamine 0.5mg/kg at a rate of 40mL over 40 minutes
- Total: Total of all reporting groups
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt | Healthy Controls | Total
Number analyzed (Participants) | 62 | 63 | 61 | 61 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 63 | 61 | 61 | 247
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.53 (11.70) | 39.94 (14.05) | 44.62 (12.26) | 37.54 (12.65) | 39.40 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 36 | 35 | 150
  Male | 26 | 20 | 25 | 26 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 60 | 62 | 59 | 60 | 241
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 1 | 2 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 11 | 13 | 47
  White | 46 | 51 | 50 | 45 | 192
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 63 | 61 | 61 | 247
Number enrolled [Count of Participants; unit: Participants] | 62 | 63 | 61 | 61 | 247

OUTCOME MEASURES:

1. Primary Outcome: Beck Scale for Suicide Ideation (BSS)
Description: The Beck Scale for Suicidal Ideation (BSSI) is a 21-item, self-report rating scale that measures the current intensity of specific attitudes, behaviors, and plans to commit suicide. Each item consists of 3 options graded according to intensity on a 3-point scale (0-2). Scores range from 0-42, with higher scores indicating more severe symptoms.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 9.09 (9.843) | 8.46 (8.954) | 1.9 (3.551)

2. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Åsberg Depression Rating Scale revised to reflect shorter timeframes will be the primary measure of change in depression. The Montgomery-Asberg Depression Rating Scale is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. A total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates mild depression, 20 to 34 indicates moderate depression, a score of 35 and greater indicates severe depression, and a total score of 60 indicates very severe depression. Scores range form 0-60, with higher scores indicating more severe symptoms.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 11.7 (10.582) | 11.56 (8.981) | 8.14 (5.338)

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The inventory contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). Anxiety symptoms are not assessed but affective, cognitive, somatic and vegetative symptoms are covered. Scoring is achieved by adding the highest ratings for all 21 items. The minimum score is 0 and maximum score is 63. Higher scores indicate greater symptom severity.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 18.02 (17.466) | 15.85 (14.641) | 12.12 (10.738)

4. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The scale is a 21-item self-report of anxiety. The total score is calculated by finding the sum of the 21 items. The scores range form 0-63, with higher scores indicating more severe symptoms.
  Score of 0 - 21 = low anxiety Score of 22 - 35 = moderate anxiety Score of 36 and above = potentially concerning levels of anxiety
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 46 | 54 | 59
units on a scale | 6.76 (10.025) | 6.59 (11.190) | 3.31 (5.240)

5. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: The Beck Hopelessness Scale is a 20-item self-report index of pessimism about the future, loss of motivation, and negative expectations. Each optimistic response is scored as 0 and each pessimistic response is scored as 1. A total score is calculated by summing the pessimistic responses for each of the 20 items. Minimum possible score is 0.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 8.25 (6.641) | 8.35 (6.253) | 7.22 (5.781)

6. Secondary Outcome: 4-item Brief Psychiatric Rating Scale (BPRS)
Description: The Brief Psychiatric Rating Scale is used to assess the presence of psychotic symptoms. This 4-item version assesses conceptual disorganization, suspiciousness/persecution, hallucinatory behavior, and unusual thought content. Each item is rated on a scale from 0 (not present) to 6 (extreme). The scores range from 0-24, with higher scores indicating more severe symptoms.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 0.02 (0.151) | 0.04 (0.272) | 0.03 (0.26)

7. Secondary Outcome: Clinician-Administered Dissociative States Scale (CADSS)
Description: The Clinician-Administered Dissociative States Scale, ascertains the presence or absence of dissociative symptoms. There are 23 clinician-administered items, each scored from 0 (not at all) to 4 (extreme). Scores range from 0-92, with higher scores indicating more severe symptoms. Items assess impairment in body sensation, perception of time and environment, memory impairment, and feelings of unreality.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 0.5 (0.902) | 0.37 (0.853) | 0.34 (0.801)

8. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: This scale assesses for manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. 13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 46 | 55 | 59
units on a scale | 1.61 (1.879) | 2.02 (3.240) | 0.85 (1.311)

9. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE)
Description: The Systematic Assessment for Treatment Emergent Events, is a 56 item, self-report inventory for adverse events. Each item is categorized by severity as: 0-none, 1-mild, 2-moderate, 3-severe. Score range is 0-168, with higher scores indicating more severe symptoms. It is designed to report adverse health events, regardless of whether or not they are suspected to be drug related, in order to reduce the under-reporting of unanticipated events compared with "known or expected" events.
  The participant numbers below correlate to the number of usable lab samples. This is the reason for discrepancy in numbers.
Time Frame: 180 minutes post dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt
Number analyzed (Participants) | 56 | 56 | 60
units on a scale | 20.66 (26.755) | 18.67 (26.36) | 11.81 (13.058)

ADVERSE EVENTS:
Time Frame: Participants were assessed for any adverse events from time of Screening visit, until after completion of Day 14 visit.
Arm/Group | MDD With Recent Suicide Attempt | MDD With Suicidal Ideation no Attempt | MDD Without Suicidal Ideation no Attempt | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/63 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 5/62 | 1/63 | 1/61 | 0/61
Other Adverse Events (participants affected / at risk) | 47/62 | 58/63 | 60/61 | 1/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDD With Recent Suicide Attempt (N=62) | MDD With Suicidal Ideation no Attempt (N=63) | MDD Without Suicidal Ideation no Attempt (N=61) | Healthy Controls (N=61)
elevated blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
worsening depression and SI (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
altered mental status (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
acute worsening depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hospitalized-worsening depression and anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hospitalized-depression,anxiety, chronic pain (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDD With Recent Suicide Attempt (N=62) | MDD With Suicidal Ideation no Attempt (N=63) | MDD Without Suicidal Ideation no Attempt (N=61) | Healthy Controls (N=61)
Dizziness (General disorders) | 13 (13) | 13 (13) | 16 (16) | 0 (0)
Numbness (Nervous system disorders) | 15 (15) | 16 (16) | 20 (20) | 0 (0)
Insomnia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 9 (9) | 9 (9) | 7 (7) | 0 (0)
Muscle or joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Myoclonus/muscle twitching (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Parasthesia/tingling (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Phantosmia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sedation (General disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Sensation needing to urinate (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin fissure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Single nightmare (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sweating (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Swelling in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 13 (13) | 9 (9) | 10 (10) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 9 (9) | 5 (5) | 0 (0)
Apathy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 6 (6) | 0 (0)
Auditory disturbance (Ear and labyrinth disorders) | 5 (5) | 3 (3) | 5 (5) | 0 (0)
Cardiovascular disturbance (Cardiac disorders) | 5 (5) | 5 (5) | 4 (4) | 1 (1)
Cold flash (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crying, tearfulness (General disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Difficulty concentrating (General disorders) | 6 (6) | 5 (5) | 7 (7) | 0 (0)
Dissociation (Psychiatric disorders) | 15 (15) | 21 (21) | 20 (20) | 0 (0)
Drowsiness,fatigue (General disorders) | 14 (14) | 17 (17) | 19 (19) | 0 (0)
Dry mouth (General disorders) | 3 (3) | 9 (9) | 4 (4) | 0 (0)
Dysgeusia (General disorders) | 7 (7) | 4 (4) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Gastrointestinal disturbance (Gastrointestinal disorders) | 8 (8) | 13 (13) | 13 (13) | 0 (0)
Hallucination (Psychiatric disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Headache (General disorders) | 3 (3) | 6 (6) | 6 (6) | 0 (0)
Hypomania (Psychiatric disorders) | 15 (15) | 10 (10) | 5 (5) | 0 (0)
Hot flash (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT02418195/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT02418195/SAP_001.pdf